CLINICAL TRIAL: NCT02027207
Title: An Individually Randomized, Placebo-controlled Trial to Measure the Protection Conferred by a Single Dose Regimen of Bivalent, Killed, Whole Cell Oral Cholera Vaccine (Shanchol™) in Dhaka, Bangladesh
Brief Title: Single Dose Oral Cholera Vaccine Study in Dhaka, Bangladesh
Acronym: SCVB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: International Vaccine Institute (Other); Government of Bangladesh (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PR-12090
Record Dates: First submitted 2013-12-23; First posted 2014-01-06 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2015-06

CONDITIONS: Cholera
Keywords: Cholera; Oral cholera vaccine; Shanchol; Protective efficacy; Bangladesh
MeSH Terms: conditions — Cholera | interventions — shanchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shanchol (Experimental)
  Interventions: Biological: Shanchol
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Shanchol — We will use the killed whole cell oral cholera vaccine, Shanchol that will be manufactured by Shantha Biotechnics, in Hyderabad, India for the study. The vaccine is registered in India and is prequalified by the WHO. Shanchol is available in a single dose vial. Vaccine will be maintained at 2-8oC. Each participant over the age of one year and non pregnant females living in communities will be individually randomized to receive vaccine.Pregnancy status will be enquired verbally for all married women of child bearing age during the census update as well as before vaccination to exclude them from the study.
  Prior to vaccination, informed consent will be taken from the adults and guardians of minor participants .Each dose of vaccine will be 1.5 ml in volume.
  Arms: Shanchol
Biological: Placebo — Placebo will be transported from the manufacturer and will be maintained at 2-8oC. Each participant over the age of one year and non pregnant females living in communities will be individually randomized to receive placebo.Each dose of placebo will be 1.5 ml in volume.Placebo will be dispensed in liquid form in identical vials.
  Arms: Placebo

SUMMARY:
Bangladesh remains endemic for cholera, which experiences biannual outbreaks with additional epidemics seen during times of floods, cyclones or any natural disaster. It affects all age groups with the majority of fatal cases occurring in children . Therefore, immunization against cholera remains an important public health component in the prevention and control of the disease .The current two-dose regimen of the internationally available oral cholera vaccines (OCV) create a logistical and programmatic challenge for use in national programs or during epidemics ,so it is important to determine if a single dose vaccine will be protective in regions where cholera is endemic. If the vaccine is found to be efficacious following a single dose, this will have profound implications for the use of the vaccine in areas with limited resources particularly in complex emergencies where a multiple dose regimen is difficult to deploy. A single-dose regimen of this vaccine will improve its 'field ability' and allow the vaccine to be used for outbreak control, especially in difficult settings where the risk of cholera is extremely high and provisions for clean water and sanitation are not available. With low OCV production rates, larger populations could be immunized against cholera if a single dose is found to be efficacious. A single-dose schedule could facilitate the inclusion of a global stockpile strategy.

The study design is a two-arm individually randomized double-blind placebo-controlled trial. The primary outcome of the study is the proportion of persons receiving 1 dose of vaccine or placebo who are detected with diarrhea with faecal excretion of V. cholera O1 in the study treatment centres from 7 days to 6 months after dosage and whose identity is confirmed through home visit.

DETAILED DESCRIPTION:
Background:

Cholera is a serious public health problem worldwide. Recently, unprecedented outbreaks have been seen in many countries including Zimbabwe, Haiti, Pakistan, Nepal, Guinea, Cuba, Congo, and Sierra Leone. These cholera outbreaks cause undue suffering with high mortality and morbidity figures as well as economic and social disruption. Bangladesh remains endemic for cholera, which peaks biannually with further increases seen during floods and cyclones .It affects all age groups, although the majority of fatal cases occur in children. Therefore, immunization against cholera remains an important public health tool for preventing and controlling the disease .

Considerable progress has been made during the last decade in the development of new generation oral vaccines against cholera. Dukoral , a killed whole cell V. cholerae O1 with recombinant B-subunit (rBS-WC), was the first to be licensed internationally and has been available mostly in developed countries as a traveller's vaccine. This vaccine is licensed in over 50 countries, including Bangladesh. The WHO now recommends Dukoral for both endemic and epidemic cholera. However, two disadvantages limit the broader use of Dukoral. First, its current price is high. Second, Dukoral needs to be administered with a buffer, which complicates large scale deployment.

The Shanchol vaccine is licensed in India and the vaccine was prequalified by the WHO in 2011.The technology for vaccine manufacturing has been transferred to Shantha Biotechnics in India (now owned by Sanofi) by IVI. A large double-blind placebo controlled phase III trial by NICED and IVI has evaluated the efficacy of the vaccine produced by Shantha in preventing diarrhea from cholera in 70,000 people in Kolkata. An analysis of the phase III trial after three years concluded that the vaccine was 66% efficacious . Advantages of the Shanchol™ vaccine include that its cost is lower and does not require administration with buffer, thus making it more feasible for use in mass vaccination programs in resource poor settings.

The current multi-dose schedules for both Dukoral and Shanchol™ have restricted the application of the oral cholera vaccine in situations where they are most needed. Getting a vaccine to the same people twice poses difficulties in the control of cholera in both endemic and epidemic settings. In a study performed in a cholera-endemic area in Kolkata, India it was found that Shanchol™ induces significant vibriocidal responses even after a single dose .This study is designed to determine the protective efficacy and duration of protection offered by a single dose regimen and is not intended to replace the recommended 2 dose regimen in endemic areas. This will be useful for epidemics and outbreaks situation.

Study population:

Mirpur has been selected for this study. Mirpur is a part of the Dhaka metropolitan area with an estimated population of over 2.5 million people. Different socio-economic groups of communities live in the area. The icddr,b hospitals treat more patients from Mirpur than from any other part of Dhaka. We have selected 9 wards in Mirpur (7-13, 15 and 41) for the study out of 16 wards. The selection has been based on the high number of cholera patients from these wards visiting the icddr,b hospitals over the last few years. Before starting the study we will commission a census of these high cholera incidence wards in Mirpur. The census team will create geographic information system (GIS) database by digitizing buildings and other structures in the target wards using satellite derived images. The digitized buildings and structures will be verified for ground verification. The census team will visit each building and ascertain whether or not people are living in the building. Based on this survey, the team will assess whether the people living in each building/structure are a high risk group or not. The census team then will collect verbal consent from the respondent and other information about the household . We will conduct a de jure census and will enumerate 324,178 high risk residents from the target wards.

Census of study population:

A paperless data collection system will be used in the census survey and subsequent census updates will also be performed biannually using handheld devices, a Samsung tab ("TAB"). The demographic surveillance will be conducted by community health workers to update the population through vital demographic events including births, deaths, internal and external migrations.

Name and description of study agents:

1. Bivalent oral killed cholera vaccine: each dose of this vaccine contains V. cholerae O1 Inaba El Tor strain Phil 6973 formalin killed 600 ELISA units (EU) of Lipopolysaccharide (LPS) V. cholerae O1 Ogawa classical strain Cairo 50 heat killed 300 EU of LPS V. cholerae O1 Ogawa classical strain Cairo 50 formalin killed 300 EU of LPS V. cholerae O1 Inaba classical strain Cairo 48 heat killed 300 EU of LPS V. cholerae O139 strain 4260B formalin killed 600 EU of LPS
2. Non Biological placebo: The composition of the placebo is as follows :

Ingredients Per 1.5 ml dose Starch: 60mg Ponceau 4R dye : 0.019 mg Brilliant blue : 0.003mg Tetrazine dye : 0.02 mg Xanthum gum : 3 mg Preservative: 0.002%(w/v)of Thiomersal (equivalent to .03 mg per 1.5 ml) Water : Up to 1.5 ml

Administration of vaccine or placebo:

The agent to be received by the participants will be determined by the randomization number on the vial. Vials will be consecutively numbered, but individually randomized into the vaccine or placebo arm. After shaking the vial properly, it will be opened and given to the participant. The contents will be poured into the mouth by the recipient, followed by intake of a small volume of water.

Census update:

The census in the study population will be updated every six months after intervention with the study agents.

Disease Surveillance:

All patients from the study area presenting for care at the hospital with diarrhea will be included in routine hospital surveillance.The diarrheal disease surveillance for the project will be conducted at icddr,b hospitals at Mohakhali and Mirpur and other health facilities for patients coming from the Mirpur study area (wards 7-13 , 15 and 41). Clinical staff at each of the two hospitals and other facilities will evaluate each patient at the hospital triage area and provide treatment as per the routine procedure.

Immunological assays using blood specimens from study participants:

Blood: Immunological analyses will be conducted in a small subgroup (334 participants) of participants .To account for unblocked unique number coding, we plan on enrolling 500 participants (less than 5 years, 5 to less than 15 years and 15 years of age or older; so as to obtain at least 108 in each age group) from the vaccination sites. Venous blood (2-5 ml) will be collected from these participants prior to immunization and 14 days after intake of the study agent.

Active follow up for safety:

We will select 6,000 participants purposively from the study participants after verbal consent is obtained. These 6,000 participants will be actively followed once every two weeks for safety outcomes for a 28 day period after study agent administration.

Primary Analysis at 6 months of follow-up:

Primary analysis will be planned at 6 months following dosing.

Analysis at 6, 12, 18 and 24 months of follow-up:

Primary analysis is to be performed at 6 months. The following available time points (12, 18 and/or 24 months will be for secondary analysis points.

Surveillance for 24 months Surveillance will be continued to complete 2 years of follow-up. Blinding will be maintained until the end of the follow-up period. The analysis at the 2 years of follow-up point will still be performed in a blinded manner.

Verbal Autopsy:

We will carry out 'Verbal Autopsy' in our study area where deaths will be identified through a household search by home visits which will be conducted by study staff. We will use two questionnaires for verbal autopsy, one for children aged 1 year to 14 years and the other for person aged 15 years and above. After identification, trained medical professional will visit homes of the deceased to perform verbal autopsy.

Pregnancy Outcome Study:

Pregnancy status in married women will be ascertained at least two months after vaccination by home visits of trained field staff. Those who will be confirmed for pregnancy at this time point will be followed up at 6 months as well as with further visits monthly to ascertain pregnancy outcome after delivery. A pregnancy follow up questionnaire will be used after consent taking for these visits

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects > 1 year of age and above Living in high risk area for cholera Provision of Informed consent for participating in the study by participant /parent or guardian as well as verbal assent for children 11-17 years.

Exclusion Criteria:

Pregnant women Aged less than 1 year History of taking cholera vaccine

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 204438 (Actual)
Dates: Start 2012-12-09 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with a single dose regimen oral cholera vaccine Shanchol will get protection | 7 days to 6 months
  Shanchol vaccine will be given to healthy, non-pregnant residents aged one and above in Dhaka, Bangladesh, against culture-proven V. cholerae O1 diarrhea which has been detected in all treatment settings serving the catchment population.

SECONDARY OUTCOMES:
Number of participants get protection with a single dose Shanchol after dosing against culture-proven V. cholerae O1 diarrhea | 7 days to 24 months
  Number of participants with a single dose Shanchol with onset of 7 days to 12 months, from 7 days to 18 months and 7 days to 24 months after dosing against culture-proven V. cholerae O1 diarrhea detected in treatment centre
Number of participants get protection with the single dose regimen of Shanchol against culture proven V. Cholerae O1 diarrhea with severe dehydration, V. Cholerae O139 diarrhea,V. Cholerae O139 diarrhea with severe dehydration . | 7 days to 24 months
  Number of participants with the single dose regimen of Shanchol against culture proven V. Cholerae O1 diarrhea with severe dehydration, V. Cholerae O139 diarrhea,V. Cholerae O139 diarrhea with severe dehydration with onset from 7 days to 12 months, from 7 days to 18 months and from 7 days to 24 months after dosing
Number of participants with a single dose Shanchol with onset of 7 days to 6 months,7 days to 12 months, from 7 days to 18 months and 7 days to 24 months after dosing against acute watery diarrhoea detected in treatment centre | 7 days to 24 months
Number of participants with a single dose Shanchol with onset of 7 days to 6 months,7 days to 12 months, from 7 days to 18 months and 7 days to 24 months after dosing against acute watery diarrhea with severe dehydration detected in treatment centre | 7 days to 24 months
Serum vibriocidal antibody responses to oral cholera vaccine Shanchol in healthy,non-pregnant residents, aged one year and older in a subset of population | 14 days
  Serum vibriocidal (To El Tor Inaba and ogawa serogroup O1 and to serogroup O139) antibody responses to a single dose regimen of the bivalent, killed, whole cell-based oral cholera vaccine Shanchol in healthy,non-pregnant residents, aged one year and older in a subset of population
Safety up to 28 days following a single dose of the bivalent, killed, whole cell oral cholera vaccine Shanchol™ administered to healthy, non-pregnant residents one year and older | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

REFERENCES:
- [Result] Kanungo S, Paisley A, Lopez AL, Bhattacharya M, Manna B, Kim DR, Han SH, Attridge S, Carbis R, Rao R, Holmgren J, Clemens JD, Sur D. Immune responses following one and two doses of the reformulated, bivalent, killed, whole-cell, oral cholera vaccine among adults and children in Kolkata, India: a randomized, placebo-controlled trial. Vaccine. 2009 Nov 16;27(49):6887-93. doi: 10.1016/j.vaccine.2009.09.008. Epub 2009 Sep 15. PMID 19761838
- [Result] Saha A, Chowdhury MI, Khanam F, Bhuiyan MS, Chowdhury F, Khan AI, Khan IA, Clemens J, Ali M, Cravioto A, Qadri F. Safety and immunogenicity study of a killed bivalent (O1 and O139) whole-cell oral cholera vaccine Shanchol, in Bangladeshi adults and children as young as 1 year of age. Vaccine. 2011 Oct 26;29(46):8285-92. doi: 10.1016/j.vaccine.2011.08.108. Epub 2011 Sep 9. PMID 21907255
- [Result] Khan IA, Saha A, Chowdhury F, Khan AI, Uddin MJ, Begum YA, Riaz BK, Islam S, Ali M, Luby SP, Clemens JD, Cravioto A, Qadri F. Coverage and cost of a large oral cholera vaccination program in a high-risk cholera endemic urban population in Dhaka, Bangladesh. Vaccine. 2013 Dec 9;31(51):6058-64. doi: 10.1016/j.vaccine.2013.10.021. Epub 2013 Oct 22. PMID 24161413
- [Derived] Chowdhury F, Bhuiyan TR, Akter A, Bhuiyan MS, Khan AI, Tauheed I, Ahmed T, Ferdous J, Dash P, Basher SR, Hakim A, Lynch J, Kim JH, Excler JL, Kim DR, Clemens JD, Qadri F. Augmented immune responses to a booster dose of oral cholera vaccine in Bangladeshi children less than 5 years of age: Revaccination after an interval of over three years of primary vaccination with a single dose of vaccine. Vaccine. 2020 Feb 11;38(7):1753-1761. doi: 10.1016/j.vaccine.2019.12.034. Epub 2019 Dec 24. PMID 31879124
- [Derived] Khan AI, Ali M, Lynch J, Kabir A, Excler JL, Khan MA, Islam MT, Akter A, Chowdhury F, Saha A, Khan IA, Desai SN, Kim DR, Saha NC, Singh AP, Clemens JD, Qadri F. Safety of a bivalent, killed, whole-cell oral cholera vaccine in pregnant women in Bangladesh: evidence from a randomized placebo-controlled trial. BMC Infect Dis. 2019 May 15;19(1):422. doi: 10.1186/s12879-019-4006-3. PMID 31092224
- [Derived] Qadri F, Ali M, Lynch J, Chowdhury F, Khan AI, Wierzba TF, Excler JL, Saha A, Islam MT, Begum YA, Bhuiyan TR, Khanam F, Chowdhury MI, Khan IA, Kabir A, Riaz BK, Akter A, Khan A, Asaduzzaman M, Kim DR, Siddik AU, Saha NC, Cravioto A, Singh AP, Clemens JD. Efficacy of a single-dose regimen of inactivated whole-cell oral cholera vaccine: results from 2 years of follow-up of a randomised trial. Lancet Infect Dis. 2018 Jun;18(6):666-674. doi: 10.1016/S1473-3099(18)30108-7. Epub 2018 Mar 14. PMID 29550406
- [Derived] Qadri F, Wierzba TF, Ali M, Chowdhury F, Khan AI, Saha A, Khan IA, Asaduzzaman M, Akter A, Khan A, Begum YA, Bhuiyan TR, Khanam F, Chowdhury MI, Islam T, Chowdhury AI, Rahman A, Siddique SA, You YA, Kim DR, Siddik AU, Saha NC, Kabir A, Cravioto A, Desai SN, Singh AP, Clemens JD. Efficacy of a Single-Dose, Inactivated Oral Cholera Vaccine in Bangladesh. N Engl J Med. 2016 May 5;374(18):1723-32. doi: 10.1056/NEJMoa1510330. PMID 27144848